CLINICAL TRIAL: NCT06334588
Title: Understanding the Mechanisms of Autism : an MRI and Social Cognition Study
Acronym: ECLAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP240105; 2023-A02668-37 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2024-02-22; First posted 2024-03-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorders; Multimodal brain imaging; Eye-tracking; Social perception; Genetics; Developmental trajectory
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Eye-Tracking Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Suspected or confirmed Autism Spectrum Disorders (ASD) (Experimental): Patient with ASD or suspected ASD for whom an MRI is requested by the clinician as part of care
  Interventions: Diagnostic Test: MRI; Device: Eye-tracking; Other: Clinical Scales; Genetic: Research of genetic anomalies
- Healthy volunteers over 3 years of age (Experimental): Healthy Control Children will be recruited specifically for the research
  Interventions: Diagnostic Test: MRI; Device: Eye-tracking; Other: Clinical Scales
- Healthy volunteers under 5 years of age (No Intervention): Children who have already undergone an MRI for various medical reasons and whose MRI was normal.

INTERVENTIONS:
Diagnostic Test: MRI — Anatomical and functional images will be acquired and review by an experienced neuro-radiologist
  Arms: Healthy volunteers over 3 years of age; Suspected or confirmed Autism Spectrum Disorders (ASD)
Device: Eye-tracking — Eye movements and follow a person's gaze will be recorded during visualization of stimuli presented in the screen by analyzing images of the eye captured by an infrared camera
  Arms: Healthy volunteers over 3 years of age; Suspected or confirmed Autism Spectrum Disorders (ASD)
Other: Clinical Scales — CGI, E-CAR and ABC will be used for behavior and clinical evaluation
  Arms: Healthy volunteers over 3 years of age; Suspected or confirmed Autism Spectrum Disorders (ASD)
Genetic: Research of genetic anomalies — For the diagnosis of autism, patients benefit from a a genetic assessment. This is carried out as part of their care
  Arms: Suspected or confirmed Autism Spectrum Disorders (ASD)

SUMMARY:
The main goal of this study is to investigate anatomo-functional brain abnormalities associated with autism spectrum disorders using a multimodal brain imaging approach, as well as its links to social cognition difficulties measured using eye-tracking

DETAILED DESCRIPTION:
Autism Spectrum Disorders (ASD) are neurodevelopmental disorders whose first manifestations appear early in childhood. Even if ASDs present a wide heterogeneity in clinical manifestations, abnormalities in social behavior, characterized in particular by a lack of preference for social information, remain the core of difficulties characteristic of autism.

Brain imaging investigations have revealed anatomo-functional abnormalities in autism, particularly in social brain regions. In parallel, eye-tracking studies have provided objective measures of social perception abnormalities in autism. These results illustrate the relevance of these research strategies in the context of ASD. Acquiring objective data on social behavior and linking them with brain imaging data opens up new avenues for research into the evolution of social skills during child development, and the brain changes underlying this process.

In this context, the main hypothesis of this study is that the investigation of the neural bases of autism spectrum disorders, using an approach combining multimodal brain imaging and the investigation of social behavior using eye-tracking, would make it possible not only to better describe abnormalities, but also to identify individual patterns at brain and behavioral level. This could help to better characterize ASDs with and without genetic abnormalities, an area which to date has received very little investigation. In addition, the objective measurements obtained with this approach would also enable the proposal of biomarkers, which would contribute not only to better monitoring of the disorder's evolution, but also to the evaluation of the effectiveness of new therapeutic interventions

ELIGIBILITY:
Inclusion Criteria:

For subjects diagnosed with ASD or suspected of ASD :

* 3 months ≤ age < 25 years ;
* an MRI required as part of the clinical procedures
* written consent obtained from parents or legal guardians.
* Affiliated to social security

For Healthy control subjects over 3 years of age:

* between 3 and 28 years of age
* no known neurological or psychiatric pathology
* written consent obtained from parents or legal guardian.
* Affiliated to social security

For Healthy control subjects under 5 years of age:

* age between 3 months and 5 years
* who have had an MRI scan in the pediatric radiology department at Necker Hospital, which was found to be normal.
* with no known neurological or psychiatric pathology
* no opposition from legal representative

Exclusion Criteria:

* Contraindication to MRI (pacemaker, intracorporeal metallic body, claustrophobia).
* Impossibility for healthy volunteers to remain still during MRI

Ages: 3 Months to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Rest cerebral blood flow (CBF) | at inclusion
  Whole brain rest CBF measured with Arterial spin labelling MRI

SECONDARY OUTCOMES:
Measurements of white matter microstructure - fractional anisotropy | at inclusion
  Measurements of white matter microstructure integrity by diffusion tensor imaging MRI, measured by fractional anisotropy (indicates the orientation of diffusion)
Measurements of white matter microstructure - mean diffusivity | at inclusion
  Measurements of white matter microstructure integrity by diffusion tensor imaging MRI, measured by mean diffusivity (the mean amount of diffusion in each of the principal directions calculated in the tensor
Measurements of white matter microstructure - radial diffusivity | at inclusion
  Measurements of white matter microstructure integrity by diffusion tensor imaging MRI, measured by radial diffusivity (the apparent water diffusion coefficient in the direction perpendicular to the axonal fibers)
Measurements of white matter microstructure - axial diffusivity | at inclusion
  Measurements of white matter microstructure integrity by diffusion tensor imaging MRI, measured by axial diffusivity (the magnitude of diffusion parallel to fiber tracts)
Measurements of resting state functional connectivity | at inclusion
  MRI-resting state measurements of correlation coefficients between different regions within different brain networks, in particular the social brain network.
Correlation between social perception and multimodal brain imaging | at inclusion
  Correlation measurements between social perception parameters measured by eye-tracking (number of fixations in social and non-social regions) and various multimodal brain imaging parameters obtained with MRI.
Correlation between clinical severity and multimodal brain imaging | at inclusion
  Measures of correlation between autism severity scores measured by the ADI-R and various multimodal brain imaging parameters obtained in MRI
Imaging abnormalities associated with known genetic mutations | at inclusion
  Multimodal brain imaging in patients with a known genetic abnormality compared with the same measures obtained in patients without known genetic abnormalities or in healthy controls.
Social perception abnormalities associated with known genetic mutations | at inclusion
  Social perception measures (number of fixations in social and non-social regions) in patients with a known genetic abnormality compared with the same measures obtained in patients without known genetic abnormalities or in healthy controls.
Anatomic changes over time - study of developmental trajectory | 2 years
  Measures of change over time (between inclusion and 2 years) in brain anatomy and function in a subgroup of ASD patients and healthy volunteers.
Social perception changes over time - study of developmental trajectory | 2 years
  Measures of change over time (between inclusion and 2 years) in social perception parameters in a subgroup of ASD patients and healthy volunteers.
Brain imaging in young children associated with ASD | at inclusion
  Multimodal brain imaging measures in young patients (<5 years) with a ASD compared with the same measures obtained in young children (<5 years) without ASD (control children)
Early data on social perception | at inclusion
  Social perception measures (number of fixations in social and non-social regions) in very young patients with ASD (3 months to 5 years) compared with a subgroup of control children aged under 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Monica ZILBOVICIUS, Study Director — INSERM INSERM ERL "Trajectoires Développementales en Psychiatrie"
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No